CLINICAL TRIAL: NCT00003447
Title: Vinorelbine Versus Gemcitabine Versus Gemcitabine and Vinorelbine in Elderly Patients With Stage IIIB-IV Non-Small Cell Lung Cancer
Brief Title: Vinorelbine and/or Gemcitabine in Treating Older Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale per lo Studio e la Cura dei Tumori (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066476; ITA-MILES; ITA-GOCSI-MILES; EU-98019
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-09

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of vinorelbine, gemcitabine, or both in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity and toxicities of gemcitabine in elderly patients with non-small cell lung cancer. II. Determine the activity and toxicity of the combination of gemcitabine and vinorelbine in these patients. III. Compare the survival rate and quality of life of these patients treated with combination chemotherapy versus single agent chemotherapy. IV. Compare objective response and time to progression of these patients treated with these chemotherapy regimens. V. Compare the toxicities of these three regimens in these patients. VI. Compare the number of hospitalizations, palliative radiation therapies, antibiotic therapies, corticosteroid therapies, analgesic therapies, and hematopoietic growth factor therapies needed for these patients treated with these chemotherapy regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, stage of disease (IIIB vs IV), and performance status (0 vs 1 vs 2). Patients are randomized to one of three treatment arms. Patients receive either vinorelbine IV, gemcitabine IV, or both on days 1 and 8 of each 21 day course. Patients who achieve an objective response or stable disease after 3 courses receive 3 more courses (for a total of 6 courses). Quality of life is assessed before treatment, after course 4 (or 3 weeks after course 3, if therapy is stopped), and at 21 days after course 6 (or 12 weeks after course 3).

PROJECTED ACCRUAL: A total of 630 patients (210 patients per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven non-small cell lung cancer Stage IV OR Stage IIIB that has supraclavicular lymph node metastases or has pleural deposits and is not curable with surgery or radical radiotherapy No brain metastases suspected clinically or demonstrated radiologically

PATIENT CHARACTERISTICS: Age: 70 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 2000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: (Unless caused by tumor) Bilirubin no greater than 1.25 times upper limit of normal (ULN) SGOT or SGPT no greater than 1.25 times ULN Renal: Creatinine no greater than 1.5 mg/dL Other: No other serious medical illness No prior or concurrent malignancy except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: No prior chemotherapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 630 (Estimated)
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, MD, Study Chair — Istituto Nazionale per lo Studio e la Cura dei Tumori
Locations (1):
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples, Italy

REFERENCES:
- [Result] Gridelli C, Perrone F, Gallo C, Cigolari S, Rossi A, Piantedosi F, Barbera S, Ferrau F, Piazza E, Rosetti F, Clerici M, Bertetto O, Robbiati SF, Frontini L, Sacco C, Castiglione F, Favaretto A, Novello S, Migliorino MR, Gasparini G, Galetta D, Iaffaioli RV, Gebbia V; MILES Investigators. Chemotherapy for elderly patients with advanced non-small-cell lung cancer: the Multicenter Italian Lung Cancer in the Elderly Study (MILES) phase III randomized trial. J Natl Cancer Inst. 2003 Mar 5;95(5):362-72. doi: 10.1093/jnci/95.5.362. PMID 12618501
- [Result] Gridelli C, Perrone S, Cigolari L, et al.: The MILES (Multicenter Italian Lung Cancer in the Elderly Study) phase 3 trial: gemcitabine + vinorelbine vs vinorelbine and vs gemcitabine in elderly advanced NSCLC patients. [Abstract] Proceedings of the American Society of Clinical Oncology A-1230, 2001.